CLINICAL TRIAL: NCT05629455
Title: CareSuperb COVID-19 Antigen Home Test Usability Study
Brief Title: CareSuperb COVID-19 Antigen Test Usability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AccessBio, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AB-1001
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is an open label study to evaluate the usability of the CareSuperb COVID-19 Antigen Home Test using information from the Quick Reference Instructions (QRI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- individuals ages 14 years and older (Experimental): This kit is intended for non-prescription home use with self-collected direct anterior nares swab samples from individuals ages 14 years and older.
  Interventions: Device: CareSuperb COVID-19 Antigen Home Test Kit
- individuals aged 2 to 13 years (Experimental): This kit is intended for non-prescription home use with self-collected direct anterior nares swab samples.
  If the subject is under the age of 14, an adult lay-user will collect the sample.
  Interventions: Device: CareSuperb COVID-19 Antigen Home Test Kit

INTERVENTIONS:
Device: CareSuperb COVID-19 Antigen Home Test Kit — At home COVID-19 antigen test kit

SUMMARY:
The purpose of this study is to evaluate the usability of the CareSuperb COVID-19 Antigen Home Test in Home Use.

DETAILED DESCRIPTION:
COVID-19 is a contagious respiratory illness, caused by infection with the novel coronavirus Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). This communicable disease is easily transmitted through aerosolized droplets containing the infectious virus. Infections with SARS-CoV-2 can have varying degrees of signs and symptoms, ranging from asymptomatic to severe. Individuals infected with SARS-CoV-2 are believed to be contagious from as early as two days prior to symptom onset to at least ten days after the onset of symptoms. The rapid detection of infections and contacts and the implementation of infection control measures are critical for mitigation of this virus.

The CareSuperb COVID-19 Antigen Home Test is a lateral flow immunochromatographic assay intended for the qualitative detection of the nucleocapsid protein antigen from SARS-CoV-2 from individuals with or without symptoms or other epidemiological reasons to suspect a COVID-19 infection. This kit is intended for non-prescription home use with self-collected direct anterior nares swab samples from individuals ages 14 years and older or adult lay user-collected anterior nares swab samples from individuals aged 2 to 13 years.

ELIGIBILITY:
Inclusion criteria:

1. An Institutional Review Board (IRB) approved informed consent / assent, if applicable, is signed and dated prior to any study-related activities.
2. Male and female subjects 2 years of age and older.
3. Subject is willing to provide a self-collected nasal swab sample. (If the subject is under the age of 14, an adult lay-user will collect the sample.)
4. Subject agrees to complete all aspects of the study.

Exclusion criteria:

1. Subject has a visual impairment that cannot be restored with glasses or contact lenses.
2. Subject has prior medical or laboratory training.
3. Subject uses home diagnostics, e.g., glucose meters, HIV tests.
4. Subject has prior knowledge of their current COVID-19 infection status.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Usability of Quick Reference Instruction | One month
  Primary Endpoints: 1. Assess the usability of the Quick Reference Instructions (QRI) based upon observer evaluation.
Usability of Test Kit | One month
  Primary Endpoints: 2. Assess the usability of the kit for home use based upon subject evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Villa, MD, Principal Investigator — L&A Morales Healthcare
Locations (1):
- L&A Morales Healthcare Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No